CLINICAL TRIAL: NCT05230719
Title: Decrease Artery Occlusion by Distal Radial Arterial Cannulation, Observational Study
Acronym: DONATION-OB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DONATION-OB
Record Dates: First submitted 2022-01-19; First posted 2022-02-09 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-01

CONDITIONS: Acute Coronary Syndrome; Procedural Complication; Outcome, Fatal
Keywords: Distal Radial Access; Radial Artery Occlusion; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Acute Coronary Syndrome; Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dTRA group: Investigators perform percutaneous coronary intervention by dTRA for patients
  Interventions: Procedure: Radial Artery Approach
- TRA group: Investigators perform percutaneous coronary intervention by conventional TRA for patients
  Interventions: Procedure: Radial Artery Approach

INTERVENTIONS:
Procedure: Radial Artery Approach — dTRA or conventional TRA for radical artery approach

SUMMARY:
The site of arterial access for coronary angiography and intervention has been the focus of research for decades as it is the source of major complications. Transradial access (TRA) reduces complications among patients undergoing percutaneous coronary procedures but is reported with the complication of radial artery occlusion (RAO) that limits the radial artery for future needs. Distal radial access (dTRA) has recently gained global popularity as an alternative access route for vascular procedures. Among the benefits of dTRA are the low risk of entry site bleeding complications, the low rate of radial artery occlusion, and improved patient and operator comfort. This study aims to reveal the feasibility and safety of dTRA and routine TRA procedures in acute coronary syndrome patients. The primary endpoints are forearm radical occlusion rate and major adverse cardiovascular events (MACEs) in the two groups. Investigators conduct this retrospected analysis to demonstrate the difference of the two procedure of Cannulation.

ELIGIBILITY:
Inclusion Criteria:

* presence of a pulse in the snuffbox

Exclusion Criteria:

* Absence of pulse
* Ultrasound indication of arterial occlusion or severe calcification
* Severe forearm artery malformation
* Patients with severe liver and renal failure, or abnormal coagulation function
* Established cardiogenic shock
* History of previous coronary artery bypass grafting and radial artery use.
* Raynaud's disease in the medical history

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the patients who received coronary angiography, based on arterial cannulation procedure, were divided into two groups, dTRA and conventional TRA. We conduct this study to illustrate the complication and MACEs of these two kinds of access.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Forearm radical | 2 years
  Doppler ultrasound to determine whether patients suffer forearm radial occlusion
MACEs | 2 years
  Major Adverse Cardiovascular Events, including cardiovascular death, myocardial infarction and heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No